CLINICAL TRIAL: NCT06408987
Title: Arthroscopically Assisted Versus Open Surgical Reduction of the Hip in Patients With Irreducible DDH Before the Walking Age
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Ebrahim Abd Allah, doctor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hip arthroscopy in DDH
Record Dates: First submitted 2024-04-15; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 .Arthroscopically assisted (Active Comparator): Arthroscopically assisted in surgical reduction of the hip in patients with irreducible DDH before the walking age arm 1
  Interventions: Procedure: arthroscopically assisted
- 2.open surgical reduction arm 2 (Active Comparator): open surgical reduction of the hip in patients with irreducible DDH before the walking age arm 2
  Interventions: Procedure: open surgical reduction

INTERVENTIONS:
Procedure: arthroscopically assisted — Arthroscopically-Assisted reduction through anterolateral portal for visualization and other accessory portals for instrumentation to achieve reduction and postoperative immobilization in a hip spica.
  Other Names: arthroscopically assisted surgical reduction
  Arms: 1 .Arthroscopically assisted
Procedure: open surgical reduction — Open reduction through a bikini incision anterior approach and postoperative immobilization in a hip spica.
  Arms: 2.open surgical reduction arm 2

SUMMARY:
To determine the role of arthroscopy in treatment of the DDH.

DETAILED DESCRIPTION:
* The term developmental dysplasia of the hip (DDH) is composed of a spectrum of pathologies from stable acetabular dysplasia (femoral head centered in acetabulum but acetabulum is shallow) to concentric hips that are unstable (femoral head can be moved in and out of the confines of the acetabulum) and frankly dislocated hips in which there is a complete loss of contact between the femoral head and acetabulum.
* Open reduction , traditionally through a Smith - Peterson approach should be considered only if closed reduction cannot be performed.
* Medial open surgical reduction is a choice for the management of patients younger than 18 months with DDH. The minimal incision and minimal blood loss are advantages of this approach. Limited exposure of the hip joint is a disadvantage.
* The arthroscopic procedure was reported to represent a meaningful alternative to the open procedure due to a lower complication rate, a safe setting, a lower rate of residual dysplasia, no observed redislocation and low rate occurrence of osteonecrosis.
* All the intra-articular structures (hypertrophic ligamentum teres, transverse acetabular ligament, and pulvinar tissue) in the acetabulum that impede the reduction of the femoral head could be eliminated by using the arthroscopic technique.

ELIGIBILITY:
* Inclusion Criteria:
* Age: - from nine months to 18 months.
* Irreducible Hip Dislocation.
* Exclusion Criteria:
* Patient age: below 9 months or above 18 months.
* Teratologic hip dislocation

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Determination the success of reduction and incidence of redislocation rate | immediately postoperative
  Documentation of concentric reduction of the hip in immediate postoperative MRI as an assessment tool for the success of the procedure.

SECONDARY OUTCOMES:
Assessment of the cosmetic appearance . | 3 month follow up
  Documentation the wound size after 3 months follow up in clinical examination as an assessment tool of cosmotic appearance
Assessment of the shortening | 1 year follow up
  Assessment the incidence of leg length discrepancy and shortening that affect walking after one year follow up in clinical examination and x-ray as an assessment tool of shortening
Assessment the incidence stiffness and decrease range of motion of the affected hip | 1 year follow up
  documentation the range of motion of the affected hip and incidence of stiffness after 6 months follow up in clinical examination as an assessment tool of stiffness.
Assessment the incidence of avascular necrosis in the affected hip | 1 year follow up
  documentation the incidence of avascular necrosis of the affected head of hip after one year follow up in clinical examination and x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Nariman aboloyoun, Ass.Prof, Study Director — Orthopedic and Trauma surgery at assiut university hospital; Hatem Galal El-Din Zaki, prof, Study Director — Orthopedic and Trauma surgery at assiut university hospital

REFERENCES:
- [Background] Roof AC, Jinguji TM, White KK. Musculoskeletal screening: developmental dysplasia of the hip. Pediatr Ann. 2013 Nov;42(11):229-35. doi: 10.3928/00904481-20131022-10. PMID 24168117
- [Background] Jenner EA, Chauhan GS, Burahee A, Choudri J, Gardner A, Bache CE. Comparison of clinical and radiological outcomes for the anterior and medial approaches to open reduction in the treatment of bilateral developmental dysplasia of the hip: a systematic review protocol. Syst Rev. 2024 Feb 23;13(1):72. doi: 10.1186/s13643-023-02444-6. PMID 38396003
- [Background] Duman S, Camurcu Y, Sofu H, Ucpunar H, Akbulut D, Yildirim T. Arthroscopic versus open, medial approach, surgical reduction for developmental dysplasia of the hip in patients under 18 months of age. Acta Orthop. 2019 Jun;90(3):292-296. doi: 10.1080/17453674.2019.1599775. Epub 2019 Apr 2. PMID 30938234
- [Background] Presch C, Eberhardt O, Wirth T, Fernandez FF. Comparison of arthroscopic and open reduction of conservatively irreducible dislocated hips of children. J Child Orthop. 2019 Aug 1;13(4):377-384. doi: 10.1302/1863-2548.13.190057. PMID 31489043
- [Background] Bulut O, Ozturk H, Tezeren G, Bulut S. Arthroscopic-assisted surgical treatment for developmental dislocation of the hip. Arthroscopy. 2005 May;21(5):574-9. doi: 10.1016/j.arthro.2005.01.004. PMID 15891724